CLINICAL TRIAL: NCT07308470
Title: Effect of Etodolac-Loaded Solid Lipid Nanoparticle Gel as an Adjunct to Physiotherapy in Knee Osteoarthritis: A Randomized Clinical Tria
Brief Title: Etodolac Nanogel as an Adjunct to Physiotherapy for Knee Osteoarthritis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pharos University in Alexandria (Other)
Responsible Party: Principal Investigator, Ola Mohamed Elsayed Elgohary, Lecturer, Department of Physical Therapy for cardiopulmonary , Pharos University, Pharos University in Alexandria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PUA-PT-ETO-KOA-2025
Record Dates: First submitted 2025-12-07; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Knee Osteoarthritis
Keywords: osteoarthritis-Etodolac
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: This is a randomized, parallel-assignment, single-blind interventional study. Thirty patients with mild to moderate unilateral knee osteoarthritis will be randomly assigned to either a control group receiving traditional physiotherapy or an experimental group receiving physiotherapy plus topical Etodolac-loaded nanoparticle gel. Outcome measures will be assessed at baseline and after 4 weeks to evaluate pain, knee function, functional performance, quadriceps strength, and proprioception
Who Masked: Outcomes Assessor
Masking Description: In this single-blind study, the outcome assessor is blinded to group allocation to minimize measurement bias. Participants and physiotherapists are aware of the treatment they receive, but all assessments of pain, knee function, functional performance, quadriceps strength, and proprioception are conducted by a blinded assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Physiotherapy + Etodolac-Loaded Nanoparticle Gel (Experimental): Participants will receive the same structured physiotherapy program as the control group, in addition to topical application of Etodolac-loaded solid lipid nanoparticle gel on the affected knee.
  Physiotherapy components:
  Quadriceps strengthening exercises
  Lower limb muscle conditioning
  Aerobic walking program
  Functional mobility exercises
  Etodolac nanogel application: Applied topically according to the study protocol to provide localized analgesic and anti-inflammatory effects.
  Duration: 4 weeks, with standardized physiotherapy sessions and daily topical gel application.
  Purpose: To evaluate whether adding Etodolac-loaded nanoparticle gel enhances pain relief, knee function, functional performance, quadriceps strength, and proprioception compared with physiotherapy alone
  Interventions: Combination Product: Etodolac-Loaded Solid Lipid Nanoparticle Gel
- Traditional Physiotherapy Exercises (Active Comparator): Participants will receive a structured physiotherapy program for knee osteoarthritis, which includes:
  Quadriceps strengthening exercises
  Lower limb muscle conditioning
  Aerobic walking program
  Functional mobility exercises
  Duration: 4 weeks, following standardized procedures for all participants. Purpose: To serve as the control group for comparison with the experimental group receiving additional Etodolac-loaded nanoparticle gel
  Interventions: Combination Product: Etodolac-Loaded Solid Lipid Nanoparticle Gel

INTERVENTIONS:
Combination Product: Etodolac-Loaded Solid Lipid Nanoparticle Gel — Physiotherapy program includes:
  Quadriceps strengthening exercises
  Lower limb muscle conditioning
  Aerobic walking program
  Functional mobility exercises
  Other Names: Traditional Aerobic Training

SUMMARY:
Brief Summary:

Knee osteoarthritis (OA) is a common, disabling condition affecting the weight-bearing knee joint, leading to pain, reduced function, and muscle weakness, particularly of the quadriceps. Strengthening exercises are recommended to improve joint stability, physical function, and slow disease progression. Etodolac, a selective NSAID approved for osteoarthritis, has proven analgesic and anti-inflammatory effects. This study investigates the adjunctive effect of a topical Etodolac-loaded solid lipid nanoparticle gel combined with traditional physiotherapy in patients with knee OA. Thirty patients with mild to moderate unilateral tibiofemoral OA will be randomized into two groups: traditional physiotherapy alone or physiotherapy plus Etodolac gel. Outcomes including pain, knee function, functional performance, quadriceps strength, and proprioception will be assessed at baseline and after four weeks. The study aims to determine whether adding topical Etodolac enhances the benefits of standard physiotherapy in managing knee OA.

DETAILED DESCRIPTION:
This randomized clinical trial investigates the effect of adding a topical Etodolac-loaded solid lipid nanoparticle gel to traditional physiotherapy in patients with mild to moderate unilateral knee osteoarthritis (OA). Thirty patients aged 45-60 years will be randomly assigned to either physiotherapy alone (control) or physiotherapy plus Etodolac nanogel (experimental) for 4 weeks. Outcomes include pain (VAS), knee function (WOMAC), functional performance (TUG, 2MWT), quadriceps strength, and proprioception. The study aims to determine whether the combination therapy provides superior pain relief, improved joint function, and enhanced muscle performance compared with physiotherapy alone, while potentially reducing systemic NSAID exposure

ELIGIBILITY:
Inclusion Criteria:

* Age between 45 and 60 years.

Mild to moderate unilateral knee osteoarthritis (Kellgren-Lawrence grades II-III).

Ability to walk independently without assistive devices.

Body Mass Index (BMI) < 30 kg/m².

No participation in resistance training in the 3 months prior to enrollment.

Referred by an orthopedic surgeon and diagnosed based on clinical and radiological examination.

Exclusion Criteria:

* Severe or bilateral knee osteoarthritis (Kellgren-Lawrence grade IV).

Congenital or acquired inflammatory, rheumatic, or neurological disorders affecting the knee.

Repeated treatment with steroids or secondary knee OA.

History of joint replacement surgery in the knee or hip.

Cardiovascular or neuromuscular disorders.

Diabetes mellitus.

Psychiatric disorders.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-08 (Estimated); Primary Completion 2026-02-07 (Estimated); Study Completion 2026-03-07 (Estimated)

PRIMARY OUTCOMES:
Pain Severity | Baseline, 4 weeks, 8 week
  Pain severity in patients with knee osteoarthritis measured using the Visual Analog Scale (VAS)Units on a 0-10 scale

SECONDARY OUTCOMES:
Functional Improvement | Baseline, 4 weeks, 8 weeks
  Improvement in knee function assessed using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) function subscale-Units on a 0-68 scale
Patient Global Assessment of Disease Activity | Baseline, 4 weeks, 8 weeks
  Patient's overall assessment of their osteoarthritis symptoms measured using a 0-100 scaleوUnits on a 0-100 scale
Physician's Global Assessmen | Baseline, 4 weeks, 8 weeks
  Physician's assessment of the patient's overall osteoarthritis status using a standardized scale-Units on a 0-100 scale

CONTACTS AND LOCATIONS:
Locations (1):
- Pharos University-Faculty of Physical Therapy, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No
Reason: Data contains sensitive patient information and will be used only for the purposes of this study under confidentiality agreements.
  Access: Data may be available upon reasonable request to the principal investigator for approved research purposes, following ethical and institutional approvals

REFERENCES:
- [Background] Trojian, T. H., Concoff, A. L., Joy, S. M., Hatzenbuehler, J. R., Saulsberry, W. J., & Coleman, C. I. (2016). AMSSM scientific statement concerning viscosupplementation injections for knee osteoarthritis: importance for individual patient outcomes. British journal of sports medicine, 50(2), 84-92. 2 Murphy, L., Schwartz, T. A., Helmick, C. G., Renner, J. B., Tudor, G., Koch, G., ... & Jordan, J. M. (2008). Lifetime risk of symptomatic knee osteoarthritis. Arthritis Care & Research, 59(9), 1207-1213. 3 Altman, R., Lim, S., Steen, R. G., & Dasa, V. (2015). Hyaluronic Acid Injections Are Associated with Delay of Total Knee Replacement Surgery in Patients with Knee Osteoarthritis: Evidence from a Large US Health Claims Database. PloS one, 10(12). 4 Jegu AG, Pereira B, Andant N, and Coudeyre E. (2014). Effect of eccentric isokinetic strengthening in the rehabilitation of patients with knee osteoarthritis: Isogo, a randomized trial. Trials; 15(1): 106. 5 Segal, N. A., Williams, G. N., Davis, M. C., Wallace, R. B., & Mikesky, A. E. (2015). Efficacy of Blood Flow-Restricted, Low-Load Resistance Training in Women with Risk Factors for Symptomatic Knee Osteoarthritis. PM&R, 7(4), 376-384